CLINICAL TRIAL: NCT02146378
Title: Vyndaqel Capsules Special Investigation -Investigation on Long-term Use-
Brief Title: Vyndaqel Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461042; NCT02146378 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Transthyretin Familial Amyloid Polyneuropathy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vyndaqel
  Interventions: Drug: Vyndaqel

INTERVENTIONS:
Drug: Vyndaqel — 20mg/day

SUMMARY:
The purpose of this study is to understand safety (e.g., occurrence of adverse drug reactions [ADRs]) and efficacy data on the long-term use of Vyndaqel Capsules (hereinafter referred to as Vyndaqel) in all patients who received this drug under actual use conditions after its marketing.

DETAILED DESCRIPTION:
Both prospective and retrospective is acceptable All the patients whom an investigator prescribes Vyndaqel should be registered

ELIGIBILITY:
Inclusion Criteria:

The subjects of this surveillance are all patients who received Vyndaqel.

Exclusion Criteria:

Patients not receive Vyndaqel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects of this surveillance are all patients who received Vyndaqel.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Konishi H, Abe H, Matsumoto N, Endo Y, Sekijima Y, Ueda M, Ando Y. Real-World Utilization Patterns, Safety, and Efficacy of Tafamidis in Patients With Hereditary Transthyretin Amyloidosis in Japan. Curr Ther Res Clin Exp. 2025 Apr 14;102:100793. doi: 10.1016/j.curtheres.2025.100793. eCollection 2025. PMID 40495907
- [Derived] Ishii T, Hirano Y, Matsumoto N, Takata A, Sekijima Y, Ueda M, Ando Y. Characteristics of Patients with Hereditary Transthyretin Amyloidosis and an Evaluation of the Safety of Tafamidis Meglumine in Japan: An Interim Analysis of an All-case Postmarketing Surveillance. Clin Ther. 2020 Sep;42(9):1728-1737.e6. doi: 10.1016/j.clinthera.2020.07.001. Epub 2020 Aug 12. PMID 32800381

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient for whom the study completed, data that might be from the same patient were combined and evaluated as the same patient, based on date of birth or age, gender, mutant genotype, name of sites that the patient visited for concomitant diseases or he/she was transferred to.
Groups:
- Vyndaqel Capsules 20mg (Tafamidis Meglumine): All of the participants who received Vyndaqel capsules 20mg as indicated in the approved local product document were observed for a period of 3 years from the start of treatment with Vyndaqel capsules 20mg (156 weeks). However, the period for participants who started to receive Vyndaqel capsules 20mg after May 2018 was 1.5 years (78 weeks). Data were collected prospectively and retrospectively.
Period: Overall Study
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Started | 402
Completed | 400
Not Completed | 2
Not completed — No information of administration | 2

BASELINE CHARACTERISTICS:
Population: A total of 500 participants were enrolled in the study, of which CRFs were collected from 494 participants. Of these 494 participants, 402 participants were determined to be included in the analysis set by data matching and identifying the same participant. Of these 402 participants (after data integration), 2 participants were excluded from the safety analysis set due to no information of administration. A total of 400 participants were included in the safety analysis set.
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 400
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 178
  ≥65 years | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 262
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ADRs in This Study
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Vyndaqel capsules 20mg in a participant who received Vyndaqel capsules 20mg.
  A serious adverse drug reaction (SADR) was ADR resulting in any of the following outcomes or deemed significant for any other reason: results in death; is life-threatening; requires inpatient hospitalization or prolongation of hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect.
  Relatedness to Vyndaqel capsules 20mg was assessed by the physician.
Time Frame: 3 years (However, the period for participants who started to receive Vyndaqel capsules 20mg after May 2018 was 1.5 years.)
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Vyndaqel capsules 20mg at least once. Participants with no information of administration were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 400
Participants
  ADR | 58
  SADR | 12

2. Secondary Outcome: Change From Baseline in the NIS-LL Score
Description: The amounts of change from baseline in the lower limbs (NIS-LL) was investigated for assessment of neurological function.The NIS-LL (Lower Limb) assessed muscle weakness, reflexes, and sensation (possible range: 0 to 88). Summary statistics at each evaluation time point and their amounts of change from the start of treatment with Vyndaqel capsules 20mg were calculated.Higher scores indicate more impaired neurological function.The mean changes from baseline in the NIS-LL at Week 78 and Week 156 were presented with standard deviation.
Time Frame: Week 78, Week 156
Population: The efficacy analysis set included participants from the safety analysis set who had at least one effectiveness evaluation by a physician based on changes in clinical symptoms and laboratory findings. Participants with non-target diseases were excluded. Among the participants in the efficacy analysis set (n=397), changes were evaluated for those with available baseline and timeframe values. The overall number of participants analyzed indicates those evaluated at week 78.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 120
Units on a scale
  Week 78 | 1.45 (4.435)
  Week 156: number analyzed (Participants) | 66
  Week 156 | 1.88 (5.620)

3. Secondary Outcome: Change From Baseline in the TQOL Score of the Norfolk QOL-DN
Description: The amounts of change from baseline in the TQOL score of the QOL-DN were used to assess quality of life .The Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) questionnaire which consists of symptoms items (1 to 7) and activities of daily living items (8 to 35) . Total Quality of Life (TQOL) (possible range: -4 to 136) in the QOL-DN was evaluated. Summary statistics at each evaluation time point and their amounts of change from the start of treatment with Vyndaqel capsules 20mg were calculated. Higher scores indicate decreased QOL.The mean changes from baseline in the TQOL score at Week 78 and Week 156 were presented with standard deviation.
Time Frame: Week 78, Week 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 122
Units on a scale
  Week 78 | 3.44 (17.043)
  Week 156: number analyzed (Participants) | 69
  Week 156 | 6.75 (24.934)

4. Secondary Outcome: Change From Baseline in mBMI
Description: Summary statistics at each evaluation time point and their amounts of change from the start of treatment with Vyndaqel capsules 20mg were calculated. Higher mBMI scores indicate better nutrition status.The mean changes from baseline in modified Body Mass Index (mBMI) at Week 26, Week 52, Week 78, Week 104, Week 130, and Week 156 were presented with standard deviation.mBMI can be calculated by multiplying BMI by the serum albumin level.In Transthyretin Familial Amyloid Polyneuropathy patients, oedema and subsequent weight gain may occur, but weight changes can be corrected with a modified BMI.
Time Frame: Week 26, Week 52, Week 78, Week 104, Week 130, Week 156
Population: The efficacy analysis set included participants from the safety analysis set who had at least one effectiveness evaluation by a physician based on changes in clinical symptoms and laboratory findings. Participants with non-target diseases were excluded. Among the participants in the efficacy analysis set (n=397), changes were evaluated for those with available baseline and timeframe values. The overall number of participants analyzed indicates those evaluated at week 26.
Measure: Mean (Standard Deviation); unit: kg/m2 x g/L
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 45
kg/m2 x g/L
  Week 26 | -6.17 (94.645)
  Week 52: number analyzed (Participants) | 32
  Week 52 | -5.63 (109.236)
  Week 78: number analyzed (Participants) | 37
  Week 78 | -28.57 (113.295)
  Week 104: number analyzed (Participants) | 15
  Week 104 | -47.26 (192.020)
  Week 130: number analyzed (Participants) | 18
  Week 130 | 11.59 (164.628)
  Week 156: number analyzed (Participants) | 16
  Week 156 | -32.81 (107.181)

5. Secondary Outcome: Time Course of Ambulatory Status
Description: The percentage of participants were calculated in each group of ambulatory status change from the start of treatment with Vyndaqel capsules 20mg to the final evaluation time point (week 156). Ambulatory status (0, 1, 2, 3a, 3b, 4) was assessed using the ambulatory ability scale. The ambulatory ability scale in the polyneuropathy dysfunction score was defined as follows. Ambulatory status 0：Walking ability is Good. Ambulatory status 1：Walking ability is able to walk without difficulty despite of sensory disorder in the lower extremities. Ambulatory status. Ambulatory status 2：Walking ability is able to walk without assistance despite of some difficulties. Ambulatory status 3a：Walking ability is able to walk with one stick or crutch. Ambulatory status 3b：Walking ability is able to walk with two sticks or crutches. Ambulatory status 4: Walking ability is unable to walk, restricted to wheelchair or bedridden.
Time Frame: Week 156
Population: The efficacy analysis set included participants from the safety analysis set who had at least one effectiveness evaluation by a physician based on changes in clinical symptoms and laboratory findings. Participants with non-target diseases were excluded. Among the participants in the efficacy analysis set (n=397), changes were evaluated for those with available baseline and week 156(n=214).
Measure: Number; unit: Percentage of Participants
Groups:
- Vyndaqel Capsules 20mg (Tafamidis Meglumine) Ambulatory Status 0: All of the participants who received Vyndaqel capsules 20mg as indicated in the approved local product document were observed for a period of 3 years from the start of treatment with Vyndaqel capsules 20mg (156 weeks). Data were collected prospectively and retrospectively.
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine) Ambulatory Status 0
Number analyzed (Participants) | 214
Percentage of Participants
  Ambulatory Status 0→0: number analyzed (Participants) | 32
  Ambulatory Status 0→0 | 15.0
  Ambulatory Status 0→1: number analyzed (Participants) | 7
  Ambulatory Status 0→1 | 3.3
  Ambulatory Status 0→2: number analyzed (Participants) | 6
  Ambulatory Status 0→2 | 2.8
  Ambulatory Status 0→3a: number analyzed (Participants) | 0
  Ambulatory Status 0→3b: number analyzed (Participants) | 1
  Ambulatory Status 0→3b | 0.5
  Ambulatory Status 0→4: number analyzed (Participants) | 1
  Ambulatory Status 0→4 | 0.5
  Ambulatory Status 0→Unconfirmed: number analyzed (Participants) | 0
  Ambulatory Status 1→0: number analyzed (Participants) | 4
  Ambulatory Status 1→0 | 1.9
  Ambulatory Status 1→1: number analyzed (Participants) | 28
  Ambulatory Status 1→1 | 13.1
  Ambulatory Status 1→2: number analyzed (Participants) | 5
  Ambulatory Status 1→2 | 2.3
  Ambulatory Status 1→3a: number analyzed (Participants) | 4
  Ambulatory Status 1→3a | 1.9
  Ambulatory Status 1→3b: number analyzed (Participants) | 0
  Ambulatory Status 1→4: number analyzed (Participants) | 2
  Ambulatory Status 1→4 | 0.9
  Ambulatory Status 1→Unconfirmed: number analyzed (Participants) | 0
  Ambulatory Status 2→0: number analyzed (Participants) | 1
  Ambulatory Status 2→0 | 0.5
  Ambulatory Status 2→1: number analyzed (Participants) | 3
  Ambulatory Status 2→1 | 1.4
  Ambulatory Status 2→2: number analyzed (Participants) | 17
  Ambulatory Status 2→2 | 7.9
  Ambulatory Status 2→3a: number analyzed (Participants) | 16
  Ambulatory Status 2→3a | 7.5
  Ambulatory Status 2→3b: number analyzed (Participants) | 8
  Ambulatory Status 2→3b | 3.7
  Ambulatory Status 2→4: number analyzed (Participants) | 12
  Ambulatory Status 2→4 | 5.6
  Ambulatory Status 2→Unconfirmed: number analyzed (Participants) | 0
  Ambulatory Status 3a→0: number analyzed (Participants) | 0
  Ambulatory Status 3a→1: number analyzed (Participants) | 1
  Ambulatory Status 3a→1 | 0.5
  Ambulatory Status 3a→2: number analyzed (Participants) | 2
  Ambulatory Status 3a→2 | 0.9
  Ambulatory Status 3a→3a: number analyzed (Participants) | 6
  Ambulatory Status 3a→3a | 2.8
  Ambulatory Status 3a→3b: number analyzed (Participants) | 2
  Ambulatory Status 3a→3b | 0.9
  Ambulatory Status 3a→4: number analyzed (Participants) | 6
  Ambulatory Status 3a→4 | 2.8
  Ambulatory Status 3a→Unconfirmed: number analyzed (Participants) | 0
  Ambulatory Status 3b→0: number analyzed (Participants) | 0
  Ambulatory Status 3b→1: number analyzed (Participants) | 0
  Ambulatory Status 3b→2: number analyzed (Participants) | 1
  Ambulatory Status 3b→2 | 0.5
  Ambulatory Status 3b→3a: number analyzed (Participants) | 1
  Ambulatory Status 3b→3a | 0.5
  Ambulatory Status 3b→3b: number analyzed (Participants) | 15
  Ambulatory Status 3b→3b | 7.0
  Ambulatory Status 3b→4: number analyzed (Participants) | 5
  Ambulatory Status 3b→4 | 2.3
  Ambulatory Status 3b→Unconfirmed: number analyzed (Participants) | 0
  Ambulatory Status 4→0: number analyzed (Participants) | 0
  Ambulatory Status 4→1: number analyzed (Participants) | 0
  Ambulatory Status 4→2: number analyzed (Participants) | 0
  Ambulatory Status 4→3a: number analyzed (Participants) | 0
  Ambulatory Status 4→3b: number analyzed (Participants) | 2
  Ambulatory Status 4→3b | 0.9
  Ambulatory Status 4→4: number analyzed (Participants) | 24
  Ambulatory Status 4→4 | 11.2
  Ambulatory Status 4→Unconfirmed: number analyzed (Participants) | 0
  Ambulatory Status Unconfirmed→0: number analyzed (Participants) | 0
  Ambulatory Status Unconfirmed→１: number analyzed (Participants) | 1
  Ambulatory Status Unconfirmed→１ | 0.5
  Ambulatory Status Unconfirmed→2: number analyzed (Participants) | 0
  Ambulatory Status Unconfirmed→3a: number analyzed (Participants) | 0
  Ambulatory Status Unconfirmed→3b: number analyzed (Participants) | 1
  Ambulatory Status Unconfirmed→3b | 0.5
  Ambulatory Status Unconfirmed→4: number analyzed (Participants) | 0
  Ambulatory Status Unconfirmed→Unconfirmed: number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in the Total Neurological Assessment Score
Description: The total score of neurological assessment (possible range: 0 to 294), scores of Motor, Reflexes and sensation were evaluated and summary statistics at each evaluation time point and their amounts of change from the start of treatment with Vyndaqel capsules 20mg were calculated. Higher scores indicate more decreased function.The mean changes from baseline in the total neurological assessment at Week 52 , Week 104, and Week 156 were presented with standard deviation.
Time Frame: Week 52, Week 104, Week 156
Population: The efficacy analysis set included participants from the safety analysis set who had at least one effectiveness evaluation by a physician based on changes in clinical symptoms and laboratory findings. Participants with non-target diseases were excluded. Among the participants in the efficacy analysis set (n=397), changes were evaluated for those with available baseline and timeframe values. The overall number of participants analyzed indicates those evaluated at week 52.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 50
Units on a scale
  Week 52 | 1.94 (7.229)
  Week 104: number analyzed (Participants) | 39
  Week 104 | 8.36 (13.927)
  Week 156: number analyzed (Participants) | 27
  Week 156 | 4.70 (11.286)

7. Secondary Outcome: Assessment of Survival Time for Death From Any Cause
Description: By setting death from any cause as events, the survival probability was estimated using the Kaplan-Meier method that treats cases who didn't have events within the observation period as censoring.
Time Frame: as for outcome 1
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation by the physician based upon change in clinical symptoms and laboratory findings at least once. Participants with non-target diseases were excluded.
Measure: Number; unit: Survival probability (%)
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 397
Survival probability (%)
  1.5y | 95.57
  3y | 87.98

8. Secondary Outcome: Assessment of Survival Time for Death Associated With ATTR-PN
Description: By setting death associated with transthyretin familial amyloid polyneuropathy (ATTR-PN) as events, the survival probability was estimated using the Kaplan-Meier method that treats cases who didn't have events within the observation period as censoring.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Number; unit: Survival probability (%)
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
Number analyzed (Participants) | 397
Survival probability (%)
  1.5y | 97.41
  3y | 94.46

ADVERSE EVENTS:
Time Frame: 3 years (However, the period for participants who started to receive Vyndaqel capsules 20mg after May 2018 was 1.5 years.)
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | Vyndaqel Capsules 20mg (Tafamidis Meglumine)
All-Cause Mortality (participants affected / at risk) | 50/400
Serious Adverse Events (participants affected / at risk) | 124/400
Other Adverse Events (participants affected / at risk) | 104/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vyndaqel Capsules 20mg (Tafamidis Meglumine) (N=400)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Atrioventricular block complete (Cardiac disorders) | 5
Atrioventricular block second degree (Cardiac disorders) | 3
Cardiac amyloidosis (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 19
Cardiac failure acute (Cardiac disorders) | 3
Cardiac failure chronic (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 2
Nodal arrhythmia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 6
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1
Visual impairment (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 4
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oesophageal stenosis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Death (General disorders) | 3
Gait disturbance (General disorders) | 2
Temperature regulation disorder (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Emphysematous cystitis (Infections and infestations) | 1
Endocarditis bacterial (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Pneumonia aspiration (Infections and infestations) | 7
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 5
Fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Autonomic neuropathy (Nervous system disorders) | 2
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 6
Dementia (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Azotaemia (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 4
Prostatitis (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 3
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vyndaqel Capsules 20mg (Tafamidis Meglumine) (N=400)
Anaemia (Blood and lymphatic system disorders) | 5
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 5
Sinus node dysfunction (Cardiac disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Ocular hypertension (Eye disorders) | 2
Retinal haemorrhage (Eye disorders) | 2
Chronic gastritis (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 9
Dysphagia (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Malaise (General disorders) | 3
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 7
Bronchitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 6
Fall (Injury, poisoning and procedural complications) | 4
Fibula fracture (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 3
Gamma-glutamyltransferase increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Carpal tunnel syndrome (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 8
Neuralgia (Nervous system disorders) | 8
Neuropathy peripheral (Nervous system disorders) | 2
Taste disorder (Nervous system disorders) | 3
Tension headache (Nervous system disorders) | 2
Hallucination (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 11
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 5
Gynaecomastia (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 3
Orthostatic hypotension (Vascular disorders) | 5
Peripheral coldness (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT02146378/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT02146378/SAP_001.pdf